CLINICAL TRIAL: NCT02284984
Title: Synergetic B-cell Immodulation in SLE
Acronym: SYNBIoSe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, YTeng, dr. Y.K.O. Teng, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL4813605814
Record Dates: First submitted 2014-10-15; First posted 2014-11-06 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Antibodies, Monoclonal; mabthera; benlysta; Antinuclear Antibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rituximab; belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab with belimumab (Experimental): Rituximab 1000mg on day 0 and day 14 Belimumab 10mg/kg on day 28, day 42 and day 56. Thereafter, patients will receive Belimumab 10mg/kg every 4 weeks.
  Interventions: Drug: Rituximab with belimumab

INTERVENTIONS:
Drug: Rituximab with belimumab — Rituximab treatment on dag 0 and 14, 1000mg iv Belimumab 10mg/kg on day 28, day 42 and day 56. Thereafter, patients will receive Belimumab 10mg/kg every 4 weeks through 72 weeks.
  Other Names: Belimumab

SUMMARY:
The present study investigates the potential of a new therapeutic approach in lupus nephritis combining rituximab (anti-CD20) and belimumab (anti-BAFF). The main goal of the study is to assess the reduction (and seroconversion) of pathogenic autoantibodies, to evaluate clinical improvement and assess the safety and feasibility of long-term B-cell depletion.

DETAILED DESCRIPTION:
Introduction Systemic lupus erythematosus (SLE) affects predominantly young women with childbearing potential (20-40 years) and inflammation can occur in virtually every organ, including kidneys, lungs, heart or brain. The disease course in SLE patients is typically characterized by frequent flares, requiring immunosuppressive treatment. Current, evidence-based treatment modalities for SLE consist of immunosuppressive treatment with high dose corticosteroids, cyclophosphamide or mycophenolic mycophenolate acid, that non-specifically target the immune system to reduce inflammation. Side-effects of these treatment strategies are (opportunistic) infections in the short term and risk for malignancy and cardiovascular disease in the long-term. Treating SLE patients with biologicals is an attractive alternative because biologicals specifically target the immune system by blocking cytokines or deplete one specific cell population, thereby reducing the risk for infections or malignancies as compared to conventional immunosuppressants. Furthermore, the scarce treatment options underscore the need to exploit new therapeutic possibilities for SLE patients who frequently experience a flare of the disease. These considerations led to the present study involving a proof-of-concept study in refractory SLE patients to assess the immunological consequences of a combination treatment with rituximab (anti-CD20) and belimumab (anti-BAFF).

Objective of the study:

A proof-of-concept study in refractory SLE patients to assess the immunological consequences of a combination treatment with rituximab (anti-CD20) and belimumab (anti-BAFF) to achieve long-term B-cell depletion. The immunological and clinical monitoring of refractory SLE patients will be monitored and the safety and feasibility of this combination treatment evaluated.

Study design:

This is a single-center, non-randomized, phase 2A, proof-of-concept study to evaluate the effects of a combination treatment with rituximab and belimumab. This combination therapy is designed to induce long-term B-cell depletion to achieve significant reduction of autoantibody-mediated immune complexes. In addition to standard therapy, SLE patients will receive 2 infusions of rituximab 1000 mg on day 0 and 14 (week 2) and belimumab on day 28 (week 4) , 42 (week 6) and 56 (week 8), then every 28 days. The primary endpoint is at 24 weeks after which an extended follow-up will take place, for subjects continuing belimumab, until 104 weeks after treatment start.

Rituximab and Belimumab will be administered intravenously according to the manufacturer's instructions. Clinical and immunological parameters will be assessed every 8-12 weeks. The study medication is not blinded for patients nor physicians. The study intends to include 15 refractory SLE patients.

Study population:

Patients with systemic lupus erythematosus, older than 18 years with refractory disease as specified by the inclusion criteria (mentioned above)

Intervention:

Rituximab Patients will be intravenously treated with Rituximab 1000mg on day 0 and day 14. Before every infusion of Rituximab patients will receive intravenous hydrocortisone 100mg together with oral acetaminophen 1000 mg and intravenous Tavegil 2 mg.

Belimumab Patients will be intravenously treated with Belimumab 10mg/kg on day 28, day 42 and day 56. Thereafter, patients will receive Belimumab 10mg/kg every 4 weeks. No pre-medication is administered

Primary study parameters/outcome of the study:

In this proof-of-concept study the primary objective is to assess whether a combination treatment of rituximab and belimumab will lead to a sustained reduction of pathogenic autoantibodies.

Secondary study parameters/outcome of the study:

The main secondary objective is to evaluate the effects of long-term B-cell depletion which will involve assessments of the clinical response correlated with immunological parameters. To this end, the relevant study parameters will be evaluated after 4 weeks (short term), 24 weeks (intermediate term) and 104 weeks (long-term).

The safety and feasibility of the combination treatment according to the WHO toxicity criteria

The clinical response of refractory SLE patients upon long-term B-cell depletion by:

* a reduction in SLEDAI scores, no new BILAG (British Isles Lupus Assessment Group) A involvement and the SLE responder index
* in case of lupus nephritis: the number of partial and complete renal responders
* the number of moderate or severe flares and renal flares

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years,
2. American College of Rheumatology (ACR) diagnosis of SLE (1997 revised criteria, see appendix 1)
3. Severe SLE flare at screening (see also section 5.2.3.2.), defined as a situation in which 1 or more of the following criteria are met:

   * Increase in SLEDAI (SLE Disease Activity Index) with 12 or more points
   * New or worse SLE-related activity of major organs, i.e.: central nervous system (CNS-) SLE (includes NPSLE), vasculitis, nephritis, pericarditis and/or myocarditis, myositis, thrombocytopenia < 60, hemolytic anemia < 4.4mmol/L (=7.0g/dL).
4. Refractory disease, defined as persisting or progressive disease activity (SLEDAI > 6 points) despite conventional immunosuppressive treatment and 1 or more of the following criteria:

   * failure of the initial induction treatment at six months, for which a switch to another induction therapy regime has already been carried out;
   * intolerance or contraindication for cyclophosphamide and mycophenolate mofetil (MMF);
   * exceeding a cumulative dose of 15 gram of cyclophosphamide;
   * a second relapse within two years after start of the initial induction therapy
   * a relative contraindication for high-dose oral or intravenous (iv) prednisone, such as avascular osteonecrosis, previous psychosis on corticosteroids, osteoporosis and/or severe obesity (BMI =35 kg/m2).
5. ANA seropositivity, as defined by a positive ANA-titer = 1:80, before and at screening :

   * Positive test results from 2 independent time points within the study screening period; OR
   * One positive historical test result and 1 positive result during the screening period. Historical documentation of a positive test of ANA (eg, ANA by HEp-2 titer, ANA by ELISA) must include the date of the test.
6. Anti-DNA seropositivity, as defined by a positive anti-dsDNA serum antibody = 30 IU/mL, before and at screening:

   * Positive test results from 2 independent time points within the study screening period.
   * One positive historical test result and 1 positive result during the screening period. Historical documentation of a positive test of anti-dsDNA (eg, anti-dsDNA by Farr assay or ELISA) must include the date of the test.
7. Immune-complex mediated complement usage, as defined by:

   * a low C3 serum level = 0.9 g/L; OR
   * a low C4 serum level = 95 mg/L; OR
   * a reduced activation of the classical pathway < 75%
8. Use of effective contraception

Exclusion Criteria:

1. Active pregnancy, as proven by a positive urine beta-HCG (human chorionic gonadotropin) test or a positive serum beta-HCG
2. Significant B-cell depletion (peripheral B-cell counts < 60x10E6)
3. Significant hypogammaglobulinemia (IgG < 8.0 g/L)
4. Immunization with a live vaccine 1 month before screening
5. Active infection at time of screening, as follows:

   * Hospitalization for treatment of infection within previous 2 months of day 0 of the study
   * Use of parenteral (intravenous of intramuscular) antibiotics ( including anti-bacterial, anti-viral, anti-fungal or anti-parasitic agents) within previous 2 months of day 0 of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Reduction of pathogenic autoantibodies | 24 weeks
  A sustained reduction of pathogenic autoantibodies, in particular anti-dsDNA autoantibodies, at 24 weeks after treatment start.

SECONDARY OUTCOMES:
Seroconversion of pathogenic autoantibodies, in particular anti-dsDNA autoantibodies | 4, 24, 104 weeks
Safety and feasibility: number of patients with (serious) adverse events | 4, 24, 104 weeks
  in accordance with the WHO toxicity criteria, including malignancy, suicidal thought/intent/behaviour
Safety and feasibility: number of patients with infectious events | 4, 24, 104 weeks
  focused on serious, Varicella-zoster virus (VZV) and opportunistic infections
Safety and feasibility: number of patients with serious hypersensitivity or infusion reactions | 4, 24, 104 weeks
Clinical response | 4, 24, 104 weeks
  * a reduction in SLEDAI scores, no new BILAG A involvement and the SLE responder index
  * in case of lupus nephritis: the number of partial and complete renal responders
  * the number of moderate or severe flares and renal flares

CONTACTS AND LOCATIONS:
Overall Officials: Onno YK Teng, MD, PhD, Principal Investigator — Leiden University Medical Center; A J Rabelink, MD, PhD, Principal Investigator — Leiden University Medical Center; T WJ Huizinga, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- LUMC, Leiden, Netherlands

REFERENCES:
- [Derived] Kraaij T, Kamerling SWA, de Rooij ENM, van Daele PLA, Bredewold OW, Bakker JA, Bajema IM, Scherer HU, Toes REM, Huizinga TJW, Rabelink TJ, van Kooten C, Teng YKO. The NET-effect of combining rituximab with belimumab in severe systemic lupus erythematosus. J Autoimmun. 2018 Jul;91:45-54. doi: 10.1016/j.jaut.2018.03.003. Epub 2018 Apr 7. PMID 29636274